CLINICAL TRIAL: NCT04950725
Title: Covid-19 Virtual Recovery Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Courtney M. Wheatley, Co-Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 21-000953
Record Dates: First submitted 2021-06-30; First posted 2021-07-06 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Covid19
Keywords: Respiratory muscle training; Covid-19; Long Hauler Syndrome; Long Covid; Nasal breathing
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Low respiratory muscle training (Experimental): Low dose of RMT and fewer repetitions and use of RMT device per week
  Interventions: Behavioral: Low dose RMT
- Respiratory muscle training for strengthening (Experimental): Higher number of sets with a slightly lower number of repetitions per set
  Interventions: Behavioral: Strength RMT
- Respiratory muscle training for strengthening and nasal breathing (Experimental): Higher number of sets with a slightly lower number of repetitions per set RMT accompanied with sets of nasal breathing
  Interventions: Behavioral: Strength RMT and nasal breathing
- Respiratory muscle training for endurance (Experimental): One set of RMT with a higher number of repetitions
  Interventions: Behavioral: Endurance RMT
- Respiratory muscle training for endurance and nasal breathing (Experimental): One set of RMT with a higher number of repetitions accompanied with sets of nasal breathing
  Interventions: Behavioral: Endurance RMT and nasal breathing

INTERVENTIONS:
Behavioral: Strength RMT — 2 sets of 10 breaths twice per day using the breather or 3 sets of 10 breaths, twice per day using the Breather Fit
  Arms: Respiratory muscle training for strengthening
Behavioral: Strength RMT and nasal breathing — 2 sets of 10 breaths twice per day using the Breather or 3 sets of 10 breaths twice per day using the Breather Fit. Subjects will also be asked to complete 2 sets of 10 nasal breathing exercises either before or after the RMT exercise.
  Arms: Respiratory muscle training for strengthening and nasal breathing
Behavioral: Endurance RMT — 15 breaths twice per day using the Breather or 20 breaths twice per day using the Breather Fit
  Arms: Respiratory muscle training for endurance
Behavioral: Endurance RMT and nasal breathing — 15 breaths twice per day using the Breather or 20 breaths twice per day using the Breather Fit at a lower intensity for a longer duration without break. Subjects will also perform 2 sets of 10 nasal breathing exercises either before or after the RMT exercise.
  Arms: Respiratory muscle training for endurance and nasal breathing
Behavioral: Low dose RMT — 10 breaths, 3 times per week, at an intensity of 3 to 4 out of 10 using the Breather device.
  Arms: Low respiratory muscle training

SUMMARY:
The purpose of this study is to determine the effects of respiratory muscle training (RMT) and nasal breathing on patients who have been infected with the SARS-CoV2 virus and continue to have lingering symptoms.

DETAILED DESCRIPTION:
This study will be conducted virtually and will be completed at home using a cell phone application. Study participation involves the use of a RMT device, and/or nasal breathing. The purpose of this research is to evaluate the impact of RMT and nasal breathing on chronic symptoms of COVID-19 in patients that have recovered from SARS-CoV2.

Subjects that have tested positive for the SARS-CoV2 infection and have completed a 14 to 30 day quarantine will be recruited.The RMT device will be used up to 2 times a day at a moderate intensity for 2 or 3 sets of 10 or 15 repetitions. Additionally, 2 sets of 10 nasal breathing techniques will be performed twice a day without the RMT device.

Subjects will complete several surveys examining symptoms, physical activity, cognitive function, and quality of life at baseline, 2 weeks, and 4 weeks. Subjects will also perform phonation (speaking/speech sounds) and sit to stand tests at baseline, 2 weeks, and 4 weeks. All data will be collected through the use of a cell phone application. The cell phone application will also provide subjects with the proper RMT protocol. Additionally, subjects will receive coaching and instructions on how to use the breathing device, as well as instructions on how to complete the phonation and sit to stand test.

ELIGIBILITY:
Inclusion criteria:

* Positive test for SARS-CoV2 within the last 3 months.
* Smartphone user.
* English speaker.
* Age 18 or above.
* US resident.

Exclusion criteria:

* Hemodynamic instability.
* Contraindications or inability to perform RMT.
* Inability to navigate study questionnaires or tasks.
* History of kidney disease, arteriosclerosis obliterans, and high calcium levels.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2268 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Change in Phonation time | change from baseline to 4 weeks
  Speaking/ speech sounds
Change in Sit to stand executions | change from baseline to 4 weeks
  How many times an individual can go from sitting to standing in one minute
Change in number of reported COVID symptoms | change from baseline to 4 weeks
  question asking to report presence of COVID-related symptoms
Change in breathing difficulty | change from baseline to 4 weeks
  rating how difficult breathing is from 1 very difficult to 5 no difficulty at all
Change in reported affect of health on physical activity | change from baseline to 4 weeks
  rating of affect from 1 affects me severely to 5 not at all affected
Change in reported cognition | change from baseline to 4 weeks
  summary score of memory, alertness, sadness, anxiety and focus getting better (1), worse (-1) or no change (0) where higher score equals more improvement

CONTACTS AND LOCATIONS:
Overall Officials: Courtney M Wheatley-Guy, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials